CLINICAL TRIAL: NCT04538157
Title: Comprehensive Geriatric Assessment for Frail Older People With Chronic Kidney Disease to Increase Attainment of Patient-Identified Goals - A Cluster Randomised Controlled Trial - The GOAL Trial
Brief Title: Comprehensive Geriatric Assessment for Frail Older People With Chronic Kidney Disease - The GOAL Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Queensland (Other)
Collaborators: National Health and Medical Research Council, Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AKTN 20.01
Record Dates: First submitted 2020-08-06; First posted 2020-09-03 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-11

CONDITIONS: Frailty; Chronic Kidney Diseases
Keywords: Goal Attainment Scaling; Frailty Index
MeSH Terms: conditions — Frailty; Renal Insufficiency, Chronic | interventions — Geriatric Assessment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comprehensive Geriatric Assessment (Experimental): Specialist co-ordinated care (known as comprehensive geriatric assessment, or CGA) was developed to address medical, social, mental health, and physical needs with the help of a skilled multi-disciplinary team.
  Interventions: Other: Comprehensive Geriatric Assessment
- Usual Care (No Intervention): Usual Care

INTERVENTIONS:
Other: Comprehensive Geriatric Assessment — A CGA is a diagnostic and therapeutic intervention which initially identifies an older person's medical, functional, psychosocial problems and then tailors coordinated management plans to address them.
  Other Names: CGA
  Arms: Comprehensive Geriatric Assessment

SUMMARY:
The GOAL trial addresses patient-prioritised research topics and outcomes and will be conducted, disseminated and implemented in partnership with patients and their caregivers. This will be the first study, internationally, to evaluate the clinical and cost effectiveness of Comprehensive Geriatric Assessment (CGA), a highly promising intervention for improving patient-important health outcomes in frail older people with Chronic Kidney Disease (CKD).

DETAILED DESCRIPTION:
There is an increasing number of frail patients with CKD, and multiple morbidities. Many of them face rapid deterioration of health, referral to residential aged care facilities and loss of independence. This substantively impairs their quality of life and has societal ramifications, including very high costs of care. Patients and carers are often overwhelmed by the multitude of decisions they have to make and may follow a care path that is in contrast to their goals.

The GOAL trial addresses patient-prioritised research topics and outcomes and will be conducted, disseminated and implemented in partnership with patients and their caregivers.

The primary objective is to test the hypothesis that in frail older people with stages 3-5 CKD, Comprehensive Geriatric Assessment (compared with usual care) will increase attainment of patient-identified goals at 3 months follow up. The secondary objectives are to test the hypotheses that the Comprehensive Geriatric Assessment will increase attainment of patient-identified goals at 6 and 12 months follow up, improve their quality of life and reduce frailty, hospital and residential aged care facility admissions while being safe and cost-effective.

In this multicentre cluster randomised controlled trial, a total of 500 adult CKD stage 3-5 patients will be recruited. Sites will be randomly allocated to either provide a Comprehensive Geriatric Assessment to participants or usual care. The primary outcome measure is goal attainment scaling at 3 months follow up. The secondary outcome measures will be goal attainment scaling at 6 and 12 months, quality of life EQ-5D-5L, frailty index, mortality, hospital and residential aged care facility admissions and cost-utility analysis.

ELIGIBILITY:
Inclusion Criteria for screening:

* Moderate to severe CKD as determined by the treating nephrologist:
* Stage 3 = eGFR 30 - 59 ml/min/1.73 m2
* Stage 4 = eGFR 15 - 29 ml/min/1.73 m2
* Stage 5/5D = eGFR below 15 ml/min/1.73m2, including patients receiving dialysis
* Aged ≥65 years, or ≥ 55 years if Aboriginal or Torres Strait Islander

For inclusion in enrolment:

* Frailty Index >0.25 (FI-CKD tool)

Exclusion Criteria:

* Estimated life expectancy of less than 12 months.
* Unable to provide informed consent and/or participate in the Goal Attainment Scaling process due to cognitive impairment or another reason.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-11-19 (Actual)

PRIMARY OUTCOMES:
Goal Attainment Scaling at 3 months | 3 months
  To determine whether CGA in frail older people with stages 3-5 CKD improves attainment of patients' own goals of care at three months.

SECONDARY OUTCOMES:
Goal Attainment Scaling at 6 and 12 months | 6 and 12 months
  To determine whether CGA improves attainments of patients' own goals of care at six and 12 months.
Quality of life using EQ-5D-5L | 3, 6 and 12 months
  To determine whether CGA improved patient's quality of life at three, six and 12 months.Quality of life will be assessed using the EQ-5D-5L
Frailty status | 3, 6 and 12 months
  To determine whether CGA favourably affects the trajectory of frailty status at three, six and 12 months. Frailty will be assessed using the Frailty Index CKD.
Mortality | 12 months
  To determine whether CGA reduces mortality during the 12 months follow-up.
Duration of hospital admissions | 12 months
  To determine whether CGA reduces the duration of hospital admissions during the 12 months follow-up.
Number of hospital admissions | 12 months
  To determine whether CGA reduces the number of hospital admissions during the 12 months follow-up.
Number of residential aged care facility admissions | 12 months
  To determine whether CGA reduces admissions to residential aged care facilities at 12 months follow-up.
Cost-effectiveness | 12 months
  Difference in the incremental cost per Quality Adjusted Life Year gained between treatment arms

OTHER OUTCOMES:
Process evaluation | 12 months
  Qualitative analysis of structured interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Hubbard, Principal Investigator — The University of Queensland
Locations (15):
- Australia (15):
  - Blacktown Hospital, Blacktown, New South Wales
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Renal Research Gosford, Gosford, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Cairns Hospital, Cairns, Queensland
  - Logan Hospital, Logan City, Queensland
  - Gold Coast Hospital, Southport, Queensland
  - Toowoomba Hospital, Toowoomba, Queensland
  - Townsville Hospital, Townsville, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Austin Health, Heidelberg, Victoria
  - Western Health, St Albans, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
  - Royal Perth Hospital, Perth, Western Australia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the primary publication, after deidentification (text, tables, figures and appendices) will be available for individual participant data meta-analysis.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 2 years and ending 5 years following main publication. Proposals may be submitted up to 5 years following article publication. After 5 years, the data will be available in our University's data warehouse but without investigator support other than deposited metadata.
Access Criteria: An independent review board will assess proposals based on the following criteria: sound science, benefit-risk balancing and research team expertise.

REFERENCES:
- [Derived] Mihala G, Hubbard RE, Logan B, Johnson DW, Viecelli AK, Forbes AB. Comprehensive geriatric assessment for frail older people with chronic kidney disease to increase attainment of patient-identified goals: Statistical analysis plan for a cluster-randomised controlled trial. Contemp Clin Trials. 2025 May;152:107881. doi: 10.1016/j.cct.2025.107881. Epub 2025 Mar 13. PMID 40089148
- [Derived] Fox ST, Hubbard R, Valks A, Matsuyama M, Kalaw E, Viecelli A, Aquino EM, Johnson D, Janda M. Protocol for the process evaluation of the GOAL trial: investigating how comprehensive geriatric assessment (CGA) improves patient-centred goal attainment in older adults with chronic kidney disease in the outpatient setting. BMJ Open. 2024 Aug 3;14(8):e076328. doi: 10.1136/bmjopen-2023-076328. PMID 39097313
- [Derived] Logan B, Viecelli AK, Johnson DW, Aquino EM, Bailey J, Comans TA, Gray LC, Hawley CM, Hickey LE, Janda M, Jaure A, Jose MD, Kalaw E, Kiriwandeniya C, Matsuyama M, Mihala G, Nguyen KH, Pascoe E, Pole JD, Polkinghorne KR, Pond D, Raj R, Reidlinger DM, Scholes-Robertson N, Varghese J, Wong G, Hubbard RE; GOAL Trial Investigators. Study protocol for The GOAL Trial: comprehensive geriatric assessment for frail older people with chronic kidney disease to increase attainment of patient-identified goals-a cluster randomised controlled trial. Trials. 2023 May 30;24(1):365. doi: 10.1186/s13063-023-07363-4. PMID 37254217